CLINICAL TRIAL: NCT01755611
Title: Bioequivalence Study Between Two Medications for Oral Administration of Minocycline in 100 mg Oral Solids in Healthy Volunteers
Brief Title: Bioequivalence Minocycline Bioequivalence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 116745
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Skin Infections (Acne)
Keywords: Minocycline; Mexico; Acne; bioequivalence
MeSH Terms: conditions — Cellulitis; Acne Vulgaris; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A(reference)/B(test) (Experimental): initial administration of reference and cross-over to test
  Interventions: Drug: Minocycline 100mg
- B(test)/A(reference) (Experimental): initial administration of test and cross-over to reference
  Interventions: Drug: Minocycline 100mg

INTERVENTIONS:
Drug: Minocycline 100mg — Test product
  Other Names: MINOPAC® is a registered trademark of LABORATORIOS DERMATOLOGICOS DARIER; S.A. DE C.V.
Drug: Minocycline 100mg — Reference product
  Other Names: MINOCIN® is a registered trademark of Wyeth Holdings Corporation

SUMMARY:
The aim of the study is to compare the bioavailability of two medications containing 100 mg of minocycline in capsules to determine bioequivalence. They are Minocycline (Minocin® is a registered trademark of Wyeth Holdings Corporation), and Minocycline (Minopac® is a registered trademark of LABORATORIOS DERMATOLOGICOS DARIER, S.A. DE C.V.). Study design is randomized, open, cross-over with two single administrations with two periods and two sequences with a wash-out period of 7 days between the periods. Subjects in the study will be 25 healthy male volunteers, 18-55 years, Blood samples will be obtained at 0.0, 0.33, 0.66, 1.0, 1.33, 1.66, 2.0, 2.33, 2.66, 3.0, 4.0, 6.0, 8.0, 12.0, 16.0, 24.0, 48.0, and 72.0 hours after medication administration in each period. Plasma minocycline levels will be determined by HPLC method with UV detection with previously validated method. Minocycline concentration data will be used to calculate Cmax, AUC0-t, and AUC0-inf with WinNonlin 5.3 software. The log transformed pharmacokinetics parameters of test and reference medications will be compared calculating ratios and 90% confidence intervals. Any adverse event will be reported.

ELIGIBILITY:
Inclusion Criteria:

Males 18-55 years. Healthy based on comprehensive medical history, lab tests, Chest x-ray, Electrocardiogram, negative tests for Hepatitis B and C, and HIV. Negative urine doping test. BMI 19-26.5 kg/m2. Lab test in normal range +/- 10%. Blood pressure 139-90/89-50, heart rate 100-55, respiratory rate 24-17, temperature 37.5-35 °C. Non-smoking at least for 10 hrs before study. Written informed consent.

Exclusion Criteria:

Hypersensitivity to study medication or other related drug. History of cardiovascular, renal, hepatic, metabolic, gastrointestinal, neurologic, endocrine, hematopoietic, psychiatric or organic condition.

Requiring any drug interfering with minocycline pharmacokinetics. Exposed to inducers or inhibitors of hepatic enzymes. Intake of possible toxic drugs 30 days before study. Intake of any drug 14 days or 7 half-lives before study. Hospitalization or severe disease 60 days before study. Receiving investigational drug out of study center 30 days before study. Blood loss or blood donation ≥ 450 ml 60 days before study. Recent history of drug abuse including alcohol. Intake of xanthine containing products 10 hrs before study. Intake of grapefruit juice or hot-spice 10 hrs before study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-06-17 (Actual); Primary Completion 2011-06-25 (Actual); Study Completion 2011-06-25 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (CMAX) of drug minocycline | 0.0, 0.33, 0.66, 1.0, 1.33, 1.66, 2.0, 2.33, 2.66, 3.0, 4.0, 6.0, 8.0, 12.0, 16.0, 24.0, 48.0, and 72.0 hours postdose
  Pharmacokinetics
Area under the plasma concentration versus time curve (AUC) of drug minocycline | 0.0, 0.33, 0.66, 1.0, 1.33, 1.66, 2.0, 2.33, 2.66, 3.0, 4.0, 6.0, 8.0, 12.0, 16.0, 24.0, 48.0, and 72.0 hours postdose
  Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- See also: Results for study 116745 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116745?search=study&search_terms=116745#rs